CLINICAL TRIAL: NCT02392858
Title: Identification, in Patients Admitted to Intensive Care for Severe Influenza Respiratory Infection, of a Predictive Biomarker of Respiratory Distress
Brief Title: Severe Influenza Cohort
Acronym: ANTIGRIPPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-A01023-44
Record Dates: First submitted 2015-03-04; First posted 2015-03-19 (Estimated); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Influenza; Severe Respiratory Infection
MeSH Terms: conditions — Influenza, Human; Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- influenza cohort (Other): Influenza is a major cause of morbidity and mortality. The investigators' first goal is to evaluate soluble HLA-G5 isoform serum level as a potential marker of greater risk of death from Influenza respiratory illness in adult and pediatric patients hospitalized in reanimation.
  1 control group of 30 patients (ancillary study) will be constitued to have reference values of the HLA-G5 marker.
  Secondly, the investigators collected respiratory samples in order to study the transcriptomic profiles of influenza-infected patients with severe symptoms.
  Interventions: Other: influenza cohort

INTERVENTIONS:
Other: influenza cohort — Influenza is a major cause of morbidity and mortality. The investigators' first goal is to evaluate soluble HLA-G5 isoform serum level as a potential marker of greater risk of death from Influenza respiratory illness in adult and pediatric patients hospitalized in reanimation. Secondly, the investigators collected respiratory samples in order to study the transcriptomic profiles of influenza-infected patients with severe symptoms.

SUMMARY:
Influenza is a major cause of morbidity and mortality. The investigators first goal is to evaluate soluble HLA-G5 isoform serum level as a potential marker of greater risk of death from Influenza respiratory illness in adult and pediatric patients hospitalized in reanimation. Secondly, the investigators collected respiratory samples in order to study the transcriptomic profiles of influenza-infected patients with severe symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patient (Adult or Pediatric)
* Hospitalized in reanimation
* With a laboratory confirmed Influenza
* That agree to take part in the study
* Affiliated to National Health Insurance

For ancillary group :

* Adult at least 60 years old
* Presenting at hospital for a blood test

Exclusion Criteria:

* non willing to participate
* Influenza infection with no respiratory symptoms
* pregnancy

For ancillary group :

* Presence of immunodepression defined by:

  * Cancer, or cancer cured for less than 2 years
  * Corticosteroids, Methotrexate (MTX), anti Tumor Necrosis Factor (TNF), anti-CD20
* Infection in progress (fever)

Ages: 1 Month to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2015-01-16 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Change in ratio of the partial pressure of oxygen in arterial blood (PaO2) to the inspired oxygen fraction (FiO2), from admission at 7 days post-admission | The first, third, fifth and seventh day of hospitalization in reanimation
  decreased arterial PaO2/FiO2 ratio ≤ 100 mmHg (≤ 13.3 kPa)

SECONDARY OUTCOMES:
All cause mortality | 90 days after hospitalization
Extracorporeal membrane oxygenation requirement | 90 days after hospitalization
SOFA score (Adult) PELOD (Pediatric) | The first, third, fifth and seventh day of hospitalization in reanimation
  Elevated Score is considered as an evidence of clinical gravity

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Sebastien CASALEGNO, MD/PhD, Principal Investigator — HOSPICES CIVILS DE LYON, Virology Department
Locations (15):
- France (15):
  - Centre de Biologie et de Pathologie Nord, Lyon, Auvergne-Rhône-Alpes
  - Hôpital Femme Mère Enfant, Bron
  - CHU service réanimation adulte, Clermont-Ferrand
  - CHU service réanimation pédiatrique, Clermont-Ferrand
  - CHU service réanimation adulte, Dijon
  - CHU service réanimation pédiatrique, Dijon
  - CHU service réanimation adulte, Grenoble
  - CHU service réanimation pédiatrique, Grenoble
  - Centre de Biologie et Pathologie Est, Lyon
  - Hôpital de la Croix Rousse-service réanimation adulte chirurgicale, Lyon
  - Hôpital de la Croix Rousse-service réanimation adulte médicale, Lyon
  - Hôpital Edouard Herriot, Lyon
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Service de Réanimation Adulte, Saint-Etienne
  - CHU Service de Réanimation Pédiatrique, Saint-Etienne

REFERENCES:
- [Result] Zhang Q, Pizzorno A, Miorin L, Bastard P, Gervais A, Le Voyer T, Bizien L, Manry J, Rosain J, Philippot Q, Goavec K, Padey B, Cupic A, Laurent E, Saker K, Vanker M, Sarekannu K; COVID Human Genetic Effort; Etablissement Francais du Sang Study Group; Constances Cohort; 3C-Dijon Study; Cerba HealthCare Group; Lyon Antigrippe Working Group; REIPI INF Working Group; Garcia-Salum T, Ferres M, Le Corre N, Sanchez-Cespedes J, Balsera-Manzanero M, Carratala J, Retamar-Gentil P, Abelenda-Alonso G, Valiente A, Tiberghien P, Zins M, Debette S, Meyts I, Haerynck F, Castagnoli R, Notarangelo LD, Gonzalez-Granado LI, Dominguez-Pinilla N, Andreakos E, Triantafyllia V, Rodriguez-Gallego C, Sole-Violan J, Ruiz-Hernandez JJ, Rodriguez de Castro F, Ferreres J, Briones M, Wauters J, Vanderbeke L, Feys S, Kuo CY, Lei WT, Ku CL, Tal G, Etzioni A, Hanna S, Fournet T, Casalegno JS, Queromes G, Argaud L, Javouhey E, Rosa-Calatrava M, Cordero E, Aydillo T, Medina RA, Kisand K, Puel A, Jouanguy E, Abel L, Cobat A, Trouillet-Assant S, Garcia-Sastre A, Casanova JL. Autoantibodies against type I IFNs in patients with critical influenza pneumonia. J Exp Med. 2022 Nov 7;219(11):e20220514. doi: 10.1084/jem.20220514. Epub 2022 Sep 16. PMID 36112363